CLINICAL TRIAL: NCT05124067
Title: Effect Of Dexmedetomidine, Dexamethasone And Ondansetron On Postoperative Nausea And Vomiting In Children Undergoing Dental Rehabilitation
Brief Title: Effect of Dexmedetomidine on Prevention of Postoperative Nausea and Vomiting in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, AHMED ABDELAZIZ SHAMA, LECTURER OF ANESTHESIA AND SURGICAL ICU, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRC13407/10/21
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Nausea and Vomiting; Post Operative Pain; Emergence Delirium
Keywords: dexmedetomidine; nausea and vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Pain, Postoperative; Emergence Delirium; Nausea; Vomiting | interventions — Dexamethasone; Ondansetron; Dexmedetomidine; Saline Solution; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Group A (DEXA) (Experimental): patients will receive dexamethasone (0.15 mg/kg IV; maximum 5 mg)
  Interventions: Drug: Dexamethasone
- Group B (ONDAN) (Experimental): patients will receive ondansetron (0.05 mg/kg IV; maximum 4 mg)
  Interventions: Drug: Ondansetron
- Group C (DEXMED) (Experimental): Patients will receive dexmedetomidine (0.3 μg/kg)
  Interventions: Drug: Dexmedetomidine
- Group D (CONTROL) (Placebo Comparator): patients will receive normal saline
  Interventions: Drug: normal Saline

INTERVENTIONS:
Drug: Dexamethasone — patients will receive dexamethasone (0.15 mg/kg IV; maximum 5 mg)
  Other Names: Dexamethasone Group
  Arms: Group A (DEXA)
Drug: Ondansetron — patients will receive ondansetron (0.05 mg/kg IV; maximum 4 mg)
  Other Names: Ondansetron Group
  Arms: Group B (ONDAN)
Drug: Dexmedetomidine — Patients will receive dexmedetomidine (0.3 μg/kg)
  Other Names: Dexmedetomidine Group
  Arms: Group C (DEXMED)
Drug: normal Saline — patients will receive normal saline.
  Other Names: Control Group
  Arms: Group D (CONTROL)

SUMMARY:
this study will aim to evaluate the effects of dexmedetomidine, dexamethasone and Ondansetron on the prevention of postoperative nausea and vomiting in children undergoing dental rehabilitation surgery.

DETAILED DESCRIPTION:
Postoperative nausea and vomiting (PONV) is one of the most common and unpleasant postoperative complications, which is a major concern in surgical patients. PONV affects about 20-40% of surgical patients, with certain high-risk patients experiencing rates of up to 80%.

It has a high incidence in children, especially for tonsillectomy and dental surgery. PONV could lead to several adverse consequences, including dehydration, electrolyte imbalance, and wound dehiscence. it has also been reported PONV is associated with delayed hospital discharge, unplanned hospital admission, and increased financial costs required for patient care.

Several anti-emetic drugs have been described for the prophylactic control of PONV. Dexamethasone is common practice in surgery, as part of a multimodal pain and antiemetic strategy.

Ondansetron is a selective 5-HT3 receptor antagonist that exhibits an anti-emetic action by antagonizing vomiting signals in the afferent pathway from the stomach or small intestine and solitary tract nucleus and is effective at preventing PONV, however, the high cost of this drug has prevented it from being widely used.

Dexmedetomidine is a highly selective α2-adrenoreceptor agonist which has been widely used in clinical practice and has been explored extensively in the pediatric population due to its beneficial effects on perioperative morbidities. In the past few years, many studies in paediatrics have been published showing that dexmedetomidine lowered postoperative pain scores and opioid consumption, decreased the incidence of emergence agitation (EA), and improved the quality of recovery in pediatric patients undergoing different surgical procedures. In addition, a small selection of studies reported that dexmedetomidine could lower the incidence of nausea or vomiting after surgery and during the use of patient-controlled analgesia (PCA) in paediatrics. However, the effect of dexmedetomidine on PONV remains poorly understood.

In this study, investigators will evaluate the effect of dexmedetomidine on preventing postoperative nausea and vomiting in children in comparison with dexamethasone and ondansetron

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients 6-12 years.
* Pediatric patients (ASA physical status I, II).
* Scheduled for dental rehabilitation surgery

Exclusion Criteria:

* Parental refusal
* Allergy or contraindication to studied medication or anaesthetic agents.
* Children with known gastroesophageal reflux disease.
* Intake of antiemetic medication within 24 hours before surgery.
* Past history or family history of previous postoperative nausea and vomiting.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-03-12 (Actual)

PRIMARY OUTCOMES:
Number of participants who will develop postoperative nausea and vomiting and rate of development | 24 hours
  Postoperative vomiting will be recorded by a nurse who will be blinded to study conditions. It will be treated if vomiting occurred more than twice in 2 minutes with granisetron (0.1mg/kg and repeated if necessary but not in less than 12 hours).

SECONDARY OUTCOMES:
Postoperative pain | 24 hours
  Postoperative pain will be assessed at 1st, 2nd, 4th, 8th, 12th, 16th and 24th hrs. Postoperative by using the Pediatric Objective Pain Scale, where each criterion scores 0 - 2 to give a total score 0 - 10, and a total score of less than 5 mean adequate analgesia
Emergence delirium | 15 minutes
  Emergence delirium using the pediatric anesthesia emergence delirium (PAED) scale at four-time points: T0: after extubation; T1: 5 min after extubation; T2: 10 min after extubation; T3: 15 min extubation.
  The PAED scale contains five items: eye contact, the purposefulness of actions, awareness of surroundings, restlessness and consolability. Each item will be scored into five grades (0-4) according to a degree, giving a maximum total of 20 points. Patients with severe agitation defined as a PAED score ≥ 10 will be treated with intravenous propofol (1 mg/kg)

OTHER OUTCOMES:
Total granisetron dose given | 24 hours
  If vomiting occurred more than twice in 2 minutes will be treated with granisetron (0.1mg/kg and repeated if necessary but not in less than 12 hours).
Number of participants with the following side effects | 24 hours
  Number of participants that will develop bradycardia, hypotension or high blood glucose

CONTACTS AND LOCATIONS:
Overall Officials: AHMED A SHAMA, MD, Principal Investigator — LECTURER OF ANESTHESIA AND SURGICAL ICU, TANTA UNIVERSITY, FACULTY OF MEDICINE; SHERIF K ARAFA, MD, Study Chair — Assistant professor of Anesthesia &ICU,Kafr El sheikh University, FACULTY OF MEDICINE; AMIR A EL-SAYED, MD, Study Chair — Assistant professor of Anesthesia &ICU,Kafr El sheikh University, FACULTY OF MEDICINE
Locations (1):
- Sharurah Armed Forces Hospital, Sharurah, Najran Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No